CLINICAL TRIAL: NCT02463357
Title: Three New Ideas to Protect Special Forces From the Stress of High Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Alma College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-0254
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Mountain Sickness
Keywords: Exercise, Aerobic; Cognitive Function
MeSH Terms: conditions — Altitude Sickness; Motor Activity | interventions — Quercetin; Methazolamide; Metformin; Nitrites

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Quercetin (Experimental): Quercetin: 500mg pill, twice daily for 5 days
  Interventions: Dietary Supplement: Quercetin
- Nifedipine+Methazolamide (Experimental): Nifedipine extended release: 30mg pill, twice daily for 5 days; Methazolamide: 125mg pill, twice daily for 5 days
  Interventions: Drug: Nifedipine extended release; Drug: Methazolamide
- Metformin (Experimental): Metformin: 500mg pill, once daily for 2 days, then 500mg twice daily at altitude (3 days)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Sugar pill manufactured to look like all other investigational products
  Interventions: Drug: Placebo
- Nitrite (Experimental): Nitrite: 20mg pill, three times daily for 5 days
  Interventions: Drug: Nitrite

INTERVENTIONS:
Dietary Supplement: Quercetin
  Arms: Quercetin
Drug: Nifedipine extended release
  Arms: Nifedipine+Methazolamide
Drug: Methazolamide
  Arms: Nifedipine+Methazolamide
Drug: Metformin
  Arms: Metformin
Drug: Placebo
  Arms: Placebo
Drug: Nitrite
  Arms: Nitrite

SUMMARY:
Acute Mountain Sickness (AMS) is a well-documented syndrome that affects 42% of non-acclimatized individuals traveling to altitudes above 10,000 feet. Decreased barometric pressure, which leads to low blood oxygen levels, is the primary casual factor of AMS. Symptoms of AMS are characterized by headache, nausea, vomiting, dizziness, fatigue and difficultly sleeping. Moreover, when people travel to high altitude, cognitive performance and endurance exercise capacity are impaired. Therefore, the goal of this research is to identify effective pharmacological agents that will help reduce the symptoms of AMS and improve physical and cognitive performance at high altitude.

The investigators will study the efficacy of the dietary supplement, quercetin, the drugs nifedipine (extended release) and methazolamide taken together, the drug metformin, and the drug nitrite in reducing symptoms of AMS and improving cognitive and exercise performance at high altitudes.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* young (18-30 years old) men who can meet APFT requirements for special operation forces (SOF) training as outlined by the US Army (42 push ups, 53 sit-ups, 6 pull-ups, 2 mile run in < 15 min 54 s)

Exclusion Criteria:

* women;
* smokers;
* participants with diseases or disorders known to be affected by hypoxia or the drugs used in this study, such as hypotension, anemia, sickle cell trait or disease, and diabetes;
* participants with a history of significant head injury, migraines or seizures;
* participants taking any medication (over-the-counter or prescription) or herbal supplements;
* participants with known flavonoid allergies;
* participants with known allergies to metformin;
* participants with known hypersensitivity reaction to nifedipine;
* participants with known allergies to sulfonamide-based drugs;
* participants with inability to be headache-free when consuming the amount of caffeine in two six ounce cups of coffee or less per day;
* exposure to high altitude above 1000m in the previous three months; or
* participants who have been on an airline flight over six hours (the lowered cabin pressure for an extended period of time approximates exposure to high altitude);
* participants who are unable to achieve the minimum physical criteria required for SOF training

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Roach, PhD, Principal Investigator — University of Colorado Anschutz Medical Campus, Altitude Research Center
Locations (1):
- Alma College, Alma, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants were excluded after consent/enrollment but prior to starting the study because some subjects did not meet baseline criteria, and others had to be excluded due to resource limitations.
Groups:
- Quercetin: Quercetin: 500mg pill, twice daily for 5 days
  Quercetin
- Nifedipine+Methazolamide: Nifedipine extended release: 30mg pill, twice daily for 5 days; Methazolamide: 125mg pill, twice daily for 5 days
  Nifedipine extended release
  Methazolamide
- Metformin: Metformin: 500mg pill, once daily for 2 days, then 500mg twice daily at altitude (3 days)
  Metformin
- Placebo: Sugar pill manufactured to look like all other investigational products
  Placebo
- Nitrite: Nitrite: 20mg pill, three times daily for 5 days
  Nitrite
Period: Overall Study
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
Started | 20 | 20 | 20 | 19 | 20
Completed | 19 | 20 | 20 | 19 | 19
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite | Total
Number analyzed (Participants) | 20 | 20 | 20 | 19 | 20 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 19 | 20 | 99
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (3.0) | 21.9 (2.6) | 21.7 (2.0) | 21.3 (1.4) | 22.0 (2.1) | 21.9 (2.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 20 | 20 | 20 | 19 | 20 | 99
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 19 | 20 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in Environmental Symptoms Questionnaire at High Altitude
Description: Self-reported assessment of AMS symptoms (headache, lightheaded, dizzy, etc.). The 11-item Environmental Symptoms Questionnaire measures Acute Mountain Sickness symptoms (nausea, weakness, lightheadedness, dizziness, headache, etc.). Possible scores range from 0 to 55 (0-5 per item), with higher scores indicating a better outcome.
Time Frame: Baseline and during high altitude exposure (3 days, AM/PM)
Population: Two participants who withdrew from the study were not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
score on a scale
  Baseline | 0.132 (0.179) | 0.122 (0.214) | 0.080 (0.132) | 0.069 (0.109) | 0.121 (0.240)
  Change at 3 days | -0.088 (0.214) | -0.073 (0.224) | 0.128 (0.425) | 0.035 (0.184) | 0.044 (0.380)

2. Primary Outcome: Change in Lake Louise AMS Scoring System at High Altitude
Description: Self-reported assessment of AMS symptoms (headache, nausea, vomiting, dizziness, fatigue and difficultly sleeping). The Lake Louise AMS Scoring System measures symptoms of altitude sickness. Possible scores range from 0 to 16, with higher scores indicating a worse outcome.
Time Frame: Baseline and during high altitude exposure (3 days, AM/PM)
Population: Two participants who withdrew from the study were not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
score on a scale
  Baseline | 0.00 (0.00) | 0.150 (0.489) | 0.150 (0.671) | 0.00 (0.00) | 0.250 (1.118)
  Change at Day 3 | 0.053 (0.229) | 0.150 (0.875) | 0.750 (2.124) | 0.632 (1.012) | 0.474 (1.896)

3. Primary Outcome: Change in Army Physical Fitness Test (APFT) at High Altitude
Description: Timed 2 mile run, push-ups, sit-ups, and pull-ups. The Army Physical Fitness Test (APFT) measures physical fitness. Higher scores indicate a better outcome. A score of 60 is considered minimum "passing" score. The maximum possible score is 300, indicating the highest level of physical fitness.
Time Frame: Baseline, 1st day at high altitude
Population: Two participants who withdrew from the study were not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
score on a scale
  Baseline | 247.2 (25.1) | 251.0 (29.4) | 254.1 (26.9) | 251.5 (23.9) | 252.1 (24.9)
  Change at Day 1 | -27.5 (23.1) | -59.2 (22.7) | -32.9 (20.5) | -23.0 (27.0) | -26.1 (20.3)

4. Primary Outcome: Change in Uphill Hike at High Altitude
Description: Timed 3.1 mile uphill run/hike, with weighted back-pack
Time Frame: 2nd day at altitude
Population: Two participants who withdrew from the study were not analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
Number analyzed (Participants) | 19 | 19 | 20 | 19 | 20
seconds | 4685 (364.4) | 4993 (595.4) | 5005 (975.9) | 4819 (685.1) | 4953 (670.5)

5. Primary Outcome: Change in Defense Automated Neurobehavioral Assessment (DANA) Reaction Time at High Altitude
Description: Battery of nine cognitive function tests. The Defense Automated Neurobehavioral Assessment (DANA) measures cognitive function and was used to measure mean reaction time. Possible scores range from 180 to 500 milliseconds, with lower scores indicating a better outcome.
Time Frame: Baseline and and 1st day at high altitude
Population: Seven participants were not analyzed due to lack of data collection at baseline.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
Number analyzed (Participants) | 17 | 19 | 19 | 17 | 18
milliseconds
  Baseline | 308.0 (34.7) | 302.2 (49.5) | 312.3 (46.1) | 333.9 (41.5) | 310.7 (29.32)
  Change from baseline at day 1 | -0.5 (27.8) | 14.2 (26.6) | -8.3 (37.9) | 0.5 (30.6) | -4.6 (30.8)

ADVERSE EVENTS:
Arm/Group | Quercetin | Nifedipine+Methazolamide | Metformin | Placebo | Nitrite
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 2/20 | 1/19 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quercetin (N=20) | Nifedipine+Methazolamide (N=20) | Metformin (N=20) | Placebo (N=19) | Nitrite (N=20)
Anxiety attack (Psychiatric disorders) | 0 (0) | NA | 1 (1) | 0 (0) | 0 (0) — Anxiety attack upon arrival at venue (participant had previous history of anxiety)
Dehydration (General disorders) | 0 (0) | NA | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | NA | 0 (0) | 1 (1) | 1 (1)
URI/ILI (Flu-like illness) (Infections and infestations) | 1 (20) | NA | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes